CLINICAL TRIAL: NCT02070939
Title: A Phase 1, Randomized, Double Blind (Sponsor Open), Placebo Controlled, Single- And Multiple Dose Escalation, Parallel Group Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-06260414 In Healthy Western And Japanese Male Subjects
Brief Title: Study To Evaluate Safety And Tolerability Of Single And Multiple Ascending Doses Of PF- 06260414 In Healthy Western And Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7411001
Record Dates: First submitted 2014-02-22; First posted 2014-02-25 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Phase 1; Randomized; Double Blind; Placebo-Controlled; Single and Multiple Dose Escalation; Safety Tolerability; PK; PD; PF-06460414
MeSH Terms: interventions — PF-06260414

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- SAD cohorts 1-7 Experimental Arm (Experimental)
  Interventions: Drug: PF-06260414
- SAD Cohorts 1-7 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- MAD cohorts 2-6 Experimental Arm (Experimental)
  Interventions: Drug: PF-06260414
- MAD cohorts 2-6 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- Japanese MAD cohort 7 Experimental arm (Experimental)
  Interventions: Drug: PF-06260414
- Japanese MAD cohort 7 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06260414 — Subjects will receive single doses of 1,3,6,30,100,200, 400 mg of PF-06260414 (solution) in a dose escalating format
  Arms: SAD cohorts 1-7 Experimental Arm
Drug: Placebo — Subjects will receive single doses of PF-06260414 matching placebo (solution) in a dose escalation format
  Arms: SAD Cohorts 1-7 Placebo Arm
Drug: PF-06260414 — Subjects will receive PF-06260414 doses (solution) twice daily for 14 days
  Arms: MAD cohorts 2-6 Experimental Arm
Drug: Placebo — Subjects will receive PF-06260414 matching placebo doses (solution) of 3, 10, 30, 100mg BID and 60 mg QD for 14 days
  Arms: MAD cohorts 2-6 Placebo Arm
Drug: PF-06260414 — Japanese subjects may receive the highest dose of PF-06460414 tested in non Japanese cohort twice daily for 14 days
  Arms: Japanese MAD cohort 7 Experimental arm
Drug: Placebo — Japanese subjects may receive PF-06260414 matching placebo doses (solution) twice daily for 14 days
  Arms: Japanese MAD cohort 7 Placebo Arm

SUMMARY:
This single and multiple ascending dose study is the first evaluation of PF-0626414, a Selective Androgen Receptor Modulator in humans. The goal is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics in healthy western and Japanese male subjects .

ELIGIBILITY:
Inclusion Criteria:

* Healthy male between the ages of 21 and 50 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Additional inclusion criteria for subjects to be enrolled in Japanese cohort only: Japanese subjects who have four Japanese grandparents born in Japan.

Exclusion Criteria:

* Serum total testosterone level <270 or >1070 ng/dL
* Serum Prostate Specific Antigen (PSA) level >4 ng/mL.
* Hematocrit >48%.
* eGFR >150 ml/min/1.73m2.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Changes from baseline vital signs (blood pressure, pulse rate, oral temperature and respiration rate) | 6 weeks
Changes from baseline in 12-lead ECG parameters | 6 weeks
  Quantitative changes in ECG intervals
Incidence and severity of treatment emergent adverse events and withdrawals due to treatment emergent adverse events | 6 weeks
Incidence and magnitude of treatment emergent clinical laboratory abnormalities including hematology (including total Hb and hematocrit), chemistry, fasting glucose, urinalysis | 6 weeks
24 hour creatinine clearance (baseline and day 14). | Baseline, Day 14
Changes from baseline in total testosterone, free testosterone, estradiol, LH, FSH, SHBG. | 6 weeks
Changes from baseline in Prostate Specific Antigen (PSA). | 6 weeks
Changes from baseline in total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides. | 6 weeks

SECONDARY OUTCOMES:
Single Dose: Cmax, Tmax, AUClast, AUCinf, CL/F, Vz/F, and t½,Cmax(dn), AUCinf(dn), AUClast(dn), t½. | 6 weeks
Multiple Dose: Cmax, Tmax Ctrough, C,av,AUC,CL/F, Vz/F, Rac , Rac,Cmax , PTR, Cmax(dn),AUCτ(dn), t½. | 6 weeks
Urinary Pharmacokinetics: Amount of PF 06260414 excreted unchanged (AE and AE%), renal clearance (CLr). | 6 weeks
Single Dose: AUC(hormone or PSA), C0(hormone or PSA), Maximum PCB, Cmax(hormone or PSA), Cmin(hormone or PSA), Tmax(hormone or PSA), Tmin(hormone or PSA). | 6 weeks
  The effects of PF- 06260414 on sex hormones (total testosterone, free testosterone, estradiol, SHBG, LH and FSH) will be evaluated according to the scheduled timepoints in single ascending dose study
Multiple Dose: AUC(hormone or PSA), C0(hormone or PSA), Cmax(hormone or PSA), Cmin(hormone or PSA), Tmax(hormone or PSA), Tmin(hormone or PSA). | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Bhattacharya I, Tarabar S, Liang Y, Pradhan V, Owens J, Oemar B. Safety, Pharmacokinetic, and Pharmacodynamic Evaluation After Single and Multiple Ascending Doses of a Novel Selective Androgen Receptor Modulator in Healthy Subjects. Clin Ther. 2016 Jun;38(6):1401-1416. doi: 10.1016/j.clinthera.2016.03.025. Epub 2016 Apr 13. PMID 27085586